CLINICAL TRIAL: NCT05933902
Title: Multicenter Retrospective Observational Study to Investigate the Characteristics and Prognosis of Patients With Acute Myocarditis in Korea
Brief Title: Multicenter Retrospective Observational Study of Acute Myocarditis in Korea
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Chonnam National University Hospital (Other); Sejong General Hospital (Other); Keimyung University Dongsan Medical Center (Other); Korea University Anam Hospital (Other); Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Hoon Yang, Professor, Samsung Medical Center
Other Study IDs: 2022-01-003-003
Record Dates: First submitted 2023-05-12; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Myocarditis Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators analyze the clinical characteristics and prognosis of patients with acute myocarditis in South Korea

DETAILED DESCRIPTION:
Acute myocarditis refers to a condition in which inflammatory cells infiltrate the heart muscle due to various causes. Until now, there is no clear treatment method for myocarditis itself, and when myocardial function deteriorates or arrhythmia occurs due to myocarditis, it is common to wait for natural recovery while performing general supportive treatment for heart failure.

Through this study, the investigators analyze the factors contributing to the long-term prognosis, myocardial recovery rate, and clinical course of myocarditis. And, the investigators plan to establish an appropriate treatment strategy necessary to increase the survival rate of patients with myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Typical myocarditis symptom and sign, such as fever, chest pain, chest discomfort or shortness of breath, accompanied by elevated myocardial enzymes
* The above condition is satisfied and additional information is obtained through imaging such as cardiac MRI or cardiac biopsy

Exclusion Criteria:

● Coronary artery disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with acute myocarditis at 6 domestic hospitals in South Korea from January 2004 to December 2021
Sampling Method: Non-Probability Sample
Enrollment: 841 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Rate of In hospital mortality | through study completion, an average of 1 year
  In hospital death by any cause

SECONDARY OUTCOMES:
Rate of all-cause mortality | through study completion, an average of 1 year
  Death by any cause during follow-up
Requirement of cardiac replacement therapy | through study completion, an average of 1 year
  Left ventricular assist device insertion or heart transplantation during follow-up
Rates of Re-hospitalization due to any cause | through study completion, an average of 1 year
  Re-hospitalization due to any cause during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Yang, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hong D, Bak M, Park H, Kim HY, Lee S, Kim IC, Hyun J, Kim SR, Kim MN, Kim KH, Yang JH. Association Between Vasoactive Inotropic Score and Clinical Outcomes in Patients With Fulminant Myocarditis. Korean Circ J. 2025 Oct;55(10):938-951. doi: 10.4070/kcj.2024.0445. Epub 2025 May 28. PMID 40628676
- [Derived] Hyun J, Pack D, Bak M, Park H, Kim HY, Lee S, Kim IC, Kim SR, Kim MN, Kim KH, Lee SE, Yang JH. Clinical Characteristics and Outcomes of Acute Myocarditis: An Analysis of Korean Multicenter Registry. Korean Circ J. 2025 May;55(5):410-422. doi: 10.4070/kcj.2024.0229. Epub 2024 Dec 10. PMID 39805629
- [Derived] Bak M, Hyun J, Park H, Kim HY, Lee S, Kim IC, Kim SR, Kim MN, Kim KH, Yang JH. Early unloading and clinical outcomes in patients with fulminant myocarditis undergoing VA-ECMO: results of a multicenter retrospective study. Rev Esp Cardiol (Engl Ed). 2025 Mar;78(3):176-184. doi: 10.1016/j.rec.2024.06.004. Epub 2024 Jun 25. English, Spanish. PMID 38936469

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT05933902/Prot_SAP_000.pdf